CLINICAL TRIAL: NCT07381881
Title: Efficacy and Efficiency of GEL-AID Gelled Water for Hydration in Institutionalized Older People
Brief Title: GEL-AID: Safe and Effective Hydration for Institutionalized Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Institut de Recerca Biomèdica de Lleida (Other); Hospital Universitari de Santa María (Lleida - Spain). (Unknown)
Responsible Party: Principal Investigator, Teresa Botigué Satorra, Doctor of Health, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI24/00413
Record Dates: First submitted 2026-01-19; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Dehydration; Urinary Infections; Respiratory Infections; Daily Fluid Intake; Mortality
Keywords: dehydration; aged; nursing homes; fluid intake; gelled water
MeSH Terms: conditions — Dehydration; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive hydration with GEL-AID.
  Interventions: Device: GEL-AID
- Control Group (Active Comparator): The control group will follow the center's standard hydration plan.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: GEL-AID — For patients with swallowing difficulties, thickened liquids with commercial thickeners and gelatin will be replaced with the GEL-AID product. The texture provided will depend on the results obtained from the Volume-Viscosity Swallow Test (V-VST). Those without swallowing difficulties will be hydrated with unmodified liquids and will also be offered GEL-AID as a replacement for gelatin.
  Arms: Intervention group
Other: Usual Care — Standard intervention. For subjects with swallowing difficulties, the hydration method will involve thickened liquids with a commercial thickener (texture adjusted according to the results obtained from the V-VST) and gelatin. Those without swallowing difficulties will be hydrated with unmodified liquids and will also be offered gelatin.
  Arms: Control Group

SUMMARY:
The objective of this clinical trial is to assess whether hydration with gelled water (GEL-AID) can improve fluid intake and reduce cases of dehydration, as well as the incidence of urinary and respiratory infections in institutionalized elderly individuals in nursing homes.

The main question this trial aims to answer is:

• Do institutionalized elderly individuals hydrated with GEL-AID increase their daily fluid intake and reduce the incidence of dehydration, urinary infections, and respiratory infections?

Participants:

The control group will follow the center's usual hydration plan. Individuals with swallowing difficulties will receive thickened liquids and/or gelatin, while those without swallowing difficulties will be hydrated with unmodified liquids or gelatin.

The intervention group will receive hydration with GEL-AID. For participants with swallowing difficulties, thickened liquids and gelatin will be replaced by GEL-AID, with texture adapted to their needs. Those without swallowing difficulties will receive unmodified liquids and GEL-AID instead of gelatin.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 65 years.

Exclusion Criteria:

* No exclusion criteria have been established.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily fluid intake | From enrollment to the end of intervention at 12 months.
  Amount in millilitres (ml)
Dehydration: Serum osmolality | Baseline and 3, 6 and 12 months
  [1,86*(Na+K)+1,15*Glucose+urea+14)] Risk dehydration ≥295 mOsm/kg Dehydration > 300mOsm/kg
Dehydration: Blood Urea Nitrogen (BUN) | Baseline and 3, 6 and 12 months
  BUN = Urea/2.1428 Dehydration > 20mg/dl
Number of urinary infections | Baseline and 3, 6 and 12 months.
  Data will be obtained through retrospective review of the clinical history
Number of respiratory infections | Baseline and 3, 6 and 12 months.
  Data will be obtained through retrospective review of the clinical history.
Mortality | Baseline and 3, 6 and 12 months.
  The number of people who will die during the study, as will be obtained from the clinical history.

SECONDARY OUTCOMES:
Current Medical Conditions | Baseline and 3, 6 and 12 months.
  Medical conditions that the participant currently has.
Pharmacological treatment | Baseline and 3, 6 and 12 months.
  Number of medications the participant takes per day and the type of each medication.
Laboratory analyses | Baseline and 3, 6 and 12 months
  Blood biochemistry and urinalysis using Combur-Test®
Efficacy and safety of swallowing | Baseline and 3, 6 and 12 months.
  Volume-Viscosity Swallow Test (V-VST): identify clinical signs of impaired efficacy (labial seal impairment, oral and pharyngeal residue, and piecemeal deglutition) and impaired safety of swallowing (voice changes, coughing, and a decrease in oxygen saturation ≥3%). It begins with nectar viscosity and progressively increases the bolus volume, then proceeds to liquid, and finally to pudding viscosity.
Nutritional status | Baseline and 3, 6 and 12 months.
  Will be assessed using the Mini Nutritional Assessment (MNA). Scores range from 0 to 30. Malnutrition will be defined as scores < 17.
Presence of lesions | Baseline and 3, 6 and 12 months.
  The number and location of lesions.
Presence of edema | Baseline and 3, 6 and 12 months.
  Yes or no
Dry skin | Baseline and 3, 6 and 12 months.
  Skin turgor: determining whether the skin remains elevated after being gently pinched and released.
Cognitive status: Mini Cognitive Examination (MEC) | Baseline and 3, 6 and 12 months.
  Values = 0 - 30. Cognitive impairment: scores <= 23
Cognitive status: Global Deterioration Scale (GDS) | Baseline and 3, 6 and 12 months.
  Values = 1 - 7. Dementia: scores ≥ 3
Functional status | Baseline and 3, 6 and 12 months.
  Barthel index. Values = 0 - 100. Functional impairment: scores < 90

OTHER OUTCOMES:
Birthdate | Baseline
  Date of birth in yyyy/mm/dd
Sex | Baseline
  Female or male sex
Marital status | Baseline
  The answer options are: single, married, in partnership (but not married), separated or divorced (currently without a partner), and wido. If the answer is "widowed," it must be specified whether the loss occurred less than one year ago or more than one year ago.
Education level | Baseline
  Choose between no formal education, primary education, secondary education, or university education.
Date of institutionalization | Baseline
  The date (yyyy/mm/dd) when the resident will be recorded as having begun institutionalization at the center.

CONTACTS AND LOCATIONS:
Locations (1):
- Residència per a la Gent Gran Lleida-Balàfia i Residència i Centre de Dia per a la Gent Gran Balàfia II, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No